CLINICAL TRIAL: NCT06750081
Title: Effect of Cross-Training on Locomotor Abilities in Children with Spastic Hemiparesis
Brief Title: Cross-Training and Locomotor Abilities in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Tamer Mohamed El-Saeed, Associate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004588
Record Dates: First submitted 2024-12-15; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Cerebral Palsy (CP); Spastic Hemiparesis
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): receive an experimental intervention
  Interventions: Other: Designed rehabilitation program
- Control (Active Comparator): another therapy used to treat the same condition
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — Exercises to improve locomotor abilities of children with CP
  Arms: Control
Other: Designed rehabilitation program — Program of exercises to enhance abilities
  Arms: Experimental

SUMMARY:
The purpose was to investigate the effect of cross-training as a method of unilateral motor priming on locomotor abilities in children with spastic unilateral cerebral palsy.

DETAILED DESCRIPTION:
Thirty children with spastic unilateral cerebral palsy were recruited from different rehabilitation centers. They were assigned randomly into two groups. Children in the control group (A) were engaged in a selected physical therapy program while those in the experimental group (B) received cross-training program followed by application of the same selected physical therapy program received by group (A). The treatment programs were conducted five times per week for six successive weeks. Measurements obtained included active ankle dorsiflexion range of motion (AROM), and the speed of walking obtained by 10-meter walking test. These measures were recorded two times: pre- and post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Spasticity grade 1 to 1+, according to the Modified Ashworth Scale.
* Can stand and walk autonomously.
* Able to follow verbal commands and instructions.

Exclusion Criteria:

* Fixed musculoskeletal deformities
* significant cognitive disorders
* significant perceptual disorders
* significant auditory disorders
* significant visual disorders

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
active ankle dorsiflexion range of motion (AROM) | Baseline and at the end - through study completion, an average of 1 year
10-meter walking test | Baseline and at the end - through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peterson MD, Lukasik L, Muth T, Esposito P, Haapala H, Gordon PM, IglayReger H, Hurvitz EA. Recumbent cross-training is a feasible and safe mode of physical activity for significantly motor-impaired adults with cerebral palsy. Arch Phys Med Rehabil. 2013 Feb;94(2):401-7. doi: 10.1016/j.apmr.2012.09.027. Epub 2012 Oct 10. PMID 23063881